CLINICAL TRIAL: NCT05562258
Title: Development and Testing of a Peer-Coaching Model for the Treatment of Eating Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Tom Hildebrandt, Professor of Psychiatry and Chief of the Division of Eating & Weight Disorders, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-22-00748
Record Dates: First submitted 2022-09-28; First posted 2022-09-30 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Eating Disorder
MeSH Terms: conditions — Feeding and Eating Disorders | interventions — Patient Education as Topic

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two conditions in a parallel design including a 12-week intervention. Participants will be recruited from the Center of Excellence in Eating and Weight Disorders Program (EWDP) until the recruitment goal of 70, 35 in each group, is reached.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Parent Coaching and Patient Education (Experimental): This group includes 12 weeks of eating disorder therapy provided to the patient. Outside of therapy, parents will have access to a coach and patients will have access to weekly educational material.
  Interventions: Behavioral: Parent Coaching and Patient Education
- Parent Education and Patient Coaching (Experimental): This group includes 12 weeks of eating disorder therapy provided to the patient. Outside of therapy, parents will have access to weekly educational material and patients will have access to a coach.
  Interventions: Behavioral: Parent Education and Patient Coaching

INTERVENTIONS:
Behavioral: Parent Coaching and Patient Education — This group includes 12 weeks of eating disorder therapy provided to the patient. Outside of therapy, parents will have access to a coach and patients will have access to weekly educational material.
  Arms: Parent Coaching and Patient Education
Behavioral: Parent Education and Patient Coaching — This group includes 12 weeks of eating disorder therapy provided to the patient. Outside of therapy, parents will have access to weekly educational material and patients will have access to a coach.
  Arms: Parent Education and Patient Coaching

SUMMARY:
This project includes developing and testing a coaching approach during the treatment of eating disorders. It is expected that with the addition of support outside of regular treatment, caregivers will experience improvements in emotional taxation and patients will strengthen skills necessary for recovery. Twelve weeks of coaching will be incorporated into standard treatment. Randomization will occur placing participants into (1) parent coaching + patient educational materials or (2) parent educational materials + patient coaching.

DETAILED DESCRIPTION:
A total of 70 adolescents with eating disorders between the ages of 12-18 and their parents/caregivers will be enrolled in a randomized-controlled trial comparing parent coaching/patient education to parent education/patient coaching. Measures will include demographics, vitals, parent and patient self-efficacy, quality of life, illness related distress/impairment, and changes in eating disorder symptoms and severity.

During a screening and consenting visit, participants will complete assessments including height, weight, demographics, and interview questions to determine inclusion/exclusion criteria and eating disorder diagnoses. At baseline, patients and parents will complete online questionnaires via a REDCap interface, measuring self-efficacy, quality of life, and illness related distress/impairment.

During the intervention, participants will attend standard therapy sessions for the treatment of eating disorders, and patients and parents will be randomized to either have access to a designated coach or weekly educational materials. Patients and parents assigned to coaching will be able to contact their coach outside of their therapy session time for 15-minute coaching calls. Completed calls will be tracked to document engagement with coaching. Patients and parents assigned to weekly education materials will receive a link, which will direct them to YouTube videos related to the skills covered in therapy for that week. They will also receive a link with a few questions to document engagement with each video.

* Coaching: A coach trained in specific skills targeted to assist in family-based therapy, will be assigned to the parent/patient to be available throughout the 12-week intervention. The coach will available between the hours of 9am - 9pm, Monday - Sunday for a brief 15-minute coaching call. During the call, the coach will remind the parent/patient of family-based skills that can be utilized in vivo to address emerging situations. If a call is running over 15 minutes, the coach will refer them to their primary therapist or emergency services.
* Educational Materials: A 2-5 minute YouTube video will be distributed to the parent/patient weekly. Videos will incorporate a new skill learned in therapy that week.

Follow-up measures will be conducted mid-way through treatment and at the end-of-treatment, and these visits will involve patients and parents repeating the assessments administered during baseline.

ELIGIBILITY:
Inclusion Criteria:

* Ages 12 to 18 at entry to the study
* DSM-5 Diagnosis of an eating disorder
* Enrollment in treatment at the Center of Excellence for Eating and Weight Disorders Speak English
* Have access to a phone with WiFi or a data plan
* Parent and child/patient both willing to participate

Exclusion Criteria:

* Current or lifetime history of learning disorder or developmental disorder
* Acute suicide risk

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in Eating Disorder Recovery Self-Efficacy Questionnaire (EDRSQ) | Baseline and 12 weeks
  Changes in patient self-efficacy will be measured using the EDRSQ, which is a 23-item instrument that assesses self-efficacy with eating disorder behaviors and attitudes. Total scores range from 1-5 with higher scores indicating greater self-efficacy. Changes in self-efficacy will be calculated using the baseline and 12-week scores from the EDRSQ.

SECONDARY OUTCOMES:
Change in Parents Versus Anorexia Scale (PVA) | Baseline and 12 weeks
  Changes in parent efficacy will be measured using the PVA which is a 7-item instrument that assesses parent's level of efficacy with helping their child with an eating disorder. Total scores range from 5-35 with higher scores indicating greater efficacy. Changes in efficacy will be calculated using the baseline and 12-week scores from the PVA.
Change in Depression Anxiety and Stress Scale (DASS) | Baseline and 12 weeks
  Changes in patient stress will be measured using the DASS. The DASS is a 42-item self-report measure of negative emotional states with subscales of depression, anxiety, and stress symptoms. Each subscale is scored 0-42, with total scores ranging from 0-126. Higher scores indicate more severe psychological distress. Changes in stress will be calculated using the baseline and 12-week total score of the DASS.
Change in Center for Epidemiologic Studies-Depression (CES-D) | Baseline and 12 weeks
  Changes in parental stress will be measured using the CES-D, which is a 20-item self-report measure evaluating depressive symptoms. Scores range from 0 to 60 with higher scores indicating greater impairment. Changes in stress will be calculated using the baseline and 12-week total score of the CES-D.
Change in the Clinical Impairment Assessment (CIA) | Baseline and 12 weeks
  Patient impairment is measured using the Clinical Impairment Assessment, which is a 16-item self-report measure of impairment from eating disorders. Responses are scored using 0, 1, 2, or 3 and the score is calculated using the sum of all items. Possible scores range between 0 - 48, with higher scores indicating more impairment and lower scores indicating less impairment. Change in impairment will be calculated using the baseline and 12-week scores from CIA.
Change in weight | Baseline and 12 weeks
  Weight will be measured in the EWDP IP clinic by study staff during all study visits. Change in weight will be calculated using the baseline and 12-week measurements.
Number of Contacts with Coach outside treatment visit | 12 weeks
  Coaching utilization will be measured by tracking the number of contacts to the coach outside of treatment visits. Utilization will be calculated using the sum of contacts throughout the 12-week treatment.
Number of Treatment visits attended | 12 weeks
  Coaching utilization will be measured by tracking the number of treatment visits attended. Utilization will be calculated using the sum of treatment visits throughout the 12-week treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Hildebrandt, PsyD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Department of Psychiatry, Eating and Weight Disorders Program, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Anonymized data can be made available upon request.